CLINICAL TRIAL: NCT06224010
Title: Respiratory Drive and Inspiratory Effort in COVID-19 Associated ARDS: a Multicentric Prospective Observational Study
Brief Title: Respiratory Drive and Inspiratory Effort in COVID-19 Associated ARDS
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Vito Fanelli MD, PhD, Associate Professor, University of Turin, Italy
Other Study IDs: CE 0084148
Record Dates: First submitted 2024-01-22; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: ARDS, Human; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; Respiratory Effort-Related Arousal; Weaning Failure; Mechanical Ventilation Complication; Acute Hypoxic Respiratory Failure
Keywords: ARDS; COVID-19; Weaning from mechanical ventilation; Respiratory drive; Inspiratory effort; Respiratory monitoring
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-COVID: * This group includes patients diagnosed with Acute Respiratory Distress Syndrome (ARDS) caused by etiologies other than COVID-19.
  * ARDS was defined following Berlin criteria (2012)
  Interventions: Other: Respiratory drive and effort assessment
- COVID-Moderate: * Moderate COVID indicates a less severe level of hypoxemia compared to the Severe COVID group (according to Berlin criteria).
  * The moderate COVID group is further characterized by a diagnosis of moderate Acute Respiratory Distress Syndrome (ARDS), based on a P/F ratio (partial pressure of oxygen/fraction of inspired oxygen) at ICU admission.
  * The diagnosis of COVID-19 in these patients was confirmed using the Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) technique.
  * RT-PCR involves collecting a sample from the lower respiratory tract and detecting the presence of SARS-CoV-2 viral RNA.
  Interventions: Other: Respiratory drive and effort assessment
- COVID-Severe: * The severe COVID group has a diagnosis of Acute Respiratory Distress Syndrome (ARDS)
  * The severity of COVID-19 in this group is determined by a P/F ratio at ICU admission, indicating a higher level of hypoxemia and a more critical clinical condition.
  * The diagnosis of COVID-19 in these patients was confirmed using the Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) technique.
  * RT-PCR involves collecting a sample from the lower respiratory tract and detecting the presence of SARS-CoV-2 viral RNA.
  Interventions: Other: Respiratory drive and effort assessment

INTERVENTIONS:
Other: Respiratory drive and effort assessment — The use of a neurally-adjusted ventilatory assist catheter, the measurement of electrical activity of the diaphragm, ∆Pocc, P0.1, and other ventilatory parameters to assess respiratory drive and effort in three cohorts of patients

SUMMARY:
Data comparing respiratory drive and effort in critically ill patients with acute respiratory distress syndrome associated to different severity of COVID-19 penumonia (CARDS) and to other risk factors are lacking. Objectives: To assess respiratory drive and effort of CARDS patients at the first transition from controlled to assisted spontaneous breathing. The second aim was the rate of a composite outcome including the need of higher level of sedation

DETAILED DESCRIPTION:
Multicenter cohort study in four Italian ICU including adults with moderate and severe CARDS (PaO2/FiO2 <100 mmHg) at ICU admission. An historical cohort of patients with ARDS from various etiologies used for comparison. Respiratory drive (P0.1), diaphragm electrical activity (EAdi), inspiratory effort derived from EAdi (∆PmusEAdi) and from deflection in airway pressure occluded (ΔPocc) (PmusΔPocc), dynamic transpulmonary driving pressure (ΔPL,dyn, the difference between peak and end-expiratory transpulmonary pressure) measured under assisted ventilation.

The main ventilatory pattern variables:

* Airway Occlusion Pressure (P0.1): Measurement of the decrease in airway pressure during an end-expiratory occlusion.
* Pmus-EAdi-derived (∆Pmus, EAdi): Measurement of the pressure generated by the respiratory muscles during inspiration derived by electrical activity of the diaphragm measurements.
* Transpulmonary pressure EAdi-derived (∆Plung,dyn): difference between peak and end-expiratory transpulmonary pressure .
* Occlusive Pressure Difference (∆Pocc): Evaluation of the pressure difference between the initial and final airway opening during inspiration.
* Pmus-∆Pocc-derived (∆Pmus, ∆Pocc): Measurement of the pressure generated by the respiratory muscles during inspiration derived by ∆Pocc (∆Pocc*0.75)
* Transpulmonary driving pressure ∆Pocc derived (∆Plung, ∆Pocc): calculated as (Peak airway pressure -PEEP) - 2/3 * ∆Pocc
* Diaphragmatic Electrical Activity (EAdi): Recording of the electrical activity of the diaphragm.
* Peak EAdi (EAdiPEAK): Determination of the highest recorded value of diaphragmatic electrical activity.
* Pressure time product of the trans-diaphragmatic pressure per breath and per minute(PTP/min): the integral of Pmusc-EAdi-derived during inspiration per breath.
* Inspiratory Delay (ID): Assessment of the time delay between the start of neural inspiration and the onset of mechanical ventilation.
* Neuro-ventilatory Efficiency (NVE): Measurement of the efficiency of the neural drive to the respiratory muscles.
* Peak Airway Opening Pressure (PawPEAK): Measurement of the peak pressure in the airway during inspiration.
* Inspiratory Pressure-Time Product (PmusEAdi/b): Calculation of the work of breathing by integrating the product of diaphragmatic electrical activity and the change in airway pressure during inspiration.
* Tidal Volume (VT): Measurement of the volume of air inspired and expired during each breath.
* Respiratory Rate: Calculation of the number of breaths per minute delivered by the mechanical ventilator.
* Inspiratory and Expiratory Time (Ti,MECH and Te,MECH): Determination of the duration of mechanical inspiration and expiration.
* Inspiratory Duty Cycle (TI/TTOT-neur): Calculation of the ratio of inspiratory time to total respiratory cycle time based on neural inspiration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of acute respiratory distress syndrome based on the Berlin criteria.
* Patients with ARDS due to confirmed COVID-19 through real-time RT-PCR on nasopharyngeal swabs or lower respiratory tract aspirates.
* Patients who had received invasive mechanical ventilation for more than 72 hours.
* Patients who were candidates for assisted ventilation.

Readiness for assisted ventilation, which was defined by the following criteria:

1. Improvement of the condition leading to acute respiratory failure.
2. Positive end-expiratory pressure lower than 10 cmH2O and inspiratory oxygen fraction lower than 0.5.
3. Richmond agitation sedation scale score between 0 and -3.
4. Ability to trigger the ventilator, i.e., decrease pressure airway opening by more than 3-4 cmH2O during a brief (5-10 seconds) end-expiratory occlusion test.

   * Hemodynamic stability without vasopressor or inotropes, except for dobutamine and norepinephrine infusion below certain thresholds (dobutamine <5 gamma/Kg/min and norepinephrine <0.3 gamma/Kg/min).
   * Normothermia.

Exclusion Criteria:

* Patients affected by neurological or neuromuscular pathology and/or known phrenic nerve dysfunction.
* Patients with any contraindication to the insertion of a nasogastric tube, such as recent upper gastrointestinal surgery or esophageal varices.
* Patients < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of acute respiratory distress syndrome due to confirmed (real-time RT-PCR on nasopharyngeal swabs, or lower respiratory tract aspirates) COVID-19 (CARDS), had received invasive mechanical ventilation for more than 72 hours and were candidates for assisted ventilation. The CARDS cohort divided into 'Moderate' and 'Severe' COVID groups according to P/F ratio at ICU admission.
  A separate cohort of patients with ARDS by etiology different from COVID-19 (No-COVID), enrolled in previous studies and with the same inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Respiratory drive | 90 breaths
  Evaluation of respiratory drive using P0.1
Neuroventilatory coupling | 90 breaths
  Evaluation of respiratory drive using EAdi PEAK
Respiratory effort | 90 breaths
  Evaluation of respiratory drive using ∆Pmus-EAdi derived, ∆Pmus-∆Pocc derived, PTP/min
Transpulmonary driving pressure | 90 breaths
  Evaluation of respiratory drive using ∆Plung, dynamic

SECONDARY OUTCOMES:
Composite outcome | within forty eight hour from assisted spontaneous breathing
  Transition from light to deep sedation (Richmond agitation sedation scale from 0/-3 to -4/-5) or from assisted to controlled ventilation within 48 hours of spontaneous assisted breathing
Intensive care unit mortality | Intensive care unit stay
  Mortality
Mortality | 60 days after measurement
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Vito Fanelli, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- S.C. Anestesia e Rianimazione 1U A.O.U.- Città della Salute e della Scienza, P.O. Molinette Corso Bramante 88-90, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Bronco A, Arrigoni Marocco S, Pozzi M, Sala V, Eronia N, Villa G, Foti G, Tagliabue G, Eger M, Pesenti A. Measurement of Diaphragmatic Electrical Activity by Surface Electromyography in Intubated Subjects and Its Relationship With Inspiratory Effort. Respir Care. 2018 Nov;63(11):1341-1349. doi: 10.4187/respcare.06176. PMID 30389829
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Background] Di Mussi R, Spadaro S, Mirabella L, Volta CA, Serio G, Staffieri F, Dambrosio M, Cinnella G, Bruno F, Grasso S. Impact of prolonged assisted ventilation on diaphragmatic efficiency: NAVA versus PSV. Crit Care. 2016 Jan 5;20:1. doi: 10.1186/s13054-015-1178-0. PMID 26728475
- [Background] Di Mussi R, Spadaro S, Volta CA, Bartolomeo N, Trerotoli P, Staffieri F, Pisani L, Iannuzziello R, Dalfino L, Murgolo F, Grasso S. Continuous assessment of neuro-ventilatory drive during 12 h of pressure support ventilation in critically ill patients. Crit Care. 2020 Nov 20;24(1):652. doi: 10.1186/s13054-020-03357-9. PMID 33218354
- [Background] Vaschetto R, Cammarota G, Colombo D, Longhini F, Grossi F, Giovanniello A, Della Corte F, Navalesi P. Effects of propofol on patient-ventilator synchrony and interaction during pressure support ventilation and neurally adjusted ventilatory assist. Crit Care Med. 2014 Jan;42(1):74-82. doi: 10.1097/CCM.0b013e31829e53dc. PMID 23982026